CLINICAL TRIAL: NCT03874676
Title: Exploration of Patient Ethics and Communication Excellence (PEACE) Rounds for Patient Care Providers: A Thematic Analysis
Brief Title: Exploration of Patient Ethics and Communication Excellence (PEACE) Rounds
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1398203
Record Dates: First submitted 2019-03-06; First posted 2019-03-14 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Resilience

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PEACE Rounds Clinicians: Nurses, physicians, care managers, chaplains, and other clinicians who attend PEACE rounds as part of their routine work in the hospital.
  Interventions: Other: PEACE Rounds

INTERVENTIONS:
Other: PEACE Rounds — PEACE Rounds are a routine process for providing self help to clinicians who care for difficult patients from the perspective of ethics and the need for cross-disciplinary communication. PEACE Rounds participants will be interviewed about how they experience the rounds and for their perspective on the effects on their own wellness and resilience.

SUMMARY:
A qualitative design using the thematic analysis method is proposed to answer the research question "What is the patient care provider's experience of PEACE rounds?" By establishing salient themes pertaining to the experience and identifying the most significant variables, the study results will also contribute to more generalizable quantitative studies. This information can be used to inform best practice in the standardization and delivery of modified PEACE Rounds.

DETAILED DESCRIPTION:
Qualitative data about participants' experiences throughout the PEACE Rounds will be collected using semi-structured interviews and participant observation. This data will be analyzed to describe and explain the perceptions that emerge from participant experience.

Qualitative Sampling Purposive samples are identified to initiate data collection and analysis, and then are used to select participants who are likely to clarify, verify, or contradict data as it is collected. Sampling concludes when the data are "saturated," which means the coded categories are well-defined and no new significant insights are emerging from additional interviews.

Semi-structured Interviews

The study team will conduct semi-structured interviews, which will be recorded and transcribed, following a consented subject's participation in at least one PEACE round. Open-ended questions, intended to elicit participants' perspectives on their experience of PEACE Rounds, will frame the interview. These are:

"What/who do you remember most vividly?" "What was most meaningful to you? "What would you change about the experience, if you could? " "Would you do it again? Why or why not?" "What, if anything, changed after PEACE rounds?"

Observation PEACE Rounds will be observed by the PI to collect data that will provide further insight to participants' experiences. Observations of interactions and reactions in real time will be documented and the data will be coded and analyzed using thematic analysis methods. Observational data will not be integrated into interview data but will be used to confirm or contrast reported data.

Qualitative Data Analysis Qualitative methodology does not seek to verify hypotheses based on logical assumptions, as quantitative measures do, instead it is used to derive salient constructs directly from the data. This methodology allows inductive understanding of participants' perceptions of their participation in PEACE Rounds.

The qualitative data will be analyzed according to the thematic analysis method based on that of Braun and Clarke . the researcher has become familiar with the data and generated an initial list of ideas that are relevant to the research objective, codes will be generated. The codes will reflect a specific feature of the data that further explicates it. After the data has been coded, the researcher will look for how different codes can be combined to create overarching themes. When there is essentially no new information coming from the codes, the data is considered saturated and no new themes are created. At this point, the researcher will review the themes and refine them, so they can be expressed in a data map expressing how they fit together to tell the story of the data.

ELIGIBILITY:
Inclusion Criteria:

1. An employee of AdventHealth (AH), or a physician with privileges there, who has participated in PEACE Rounds at AdventHealth.
2. Over the age of 18
3. Able to provide informed consent
4. Must speak and understand English

Exclusion Criteria:

1. Discernable cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An employee of AdventHealth (AH), or a physician with privileges there, who has participated in PEACE Rounds at AdventHealth. This includes nurses, technicians, chaplains, care managers, child life specialists, and other clinical staff who may provide services or treatment to patients who are the subject of PEACE Rounds.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Thematic Analysis of Interview Data to Describe Effects of PEACE Rounds on Burnout Relief | 6 months
  Analysis of data collected throughout the study, using saturation sampling and documented coding techniques, will result in thematic descriptions of the aggregated experiences of clinical staff who participate in PEACE rounds. Semi-structured interviews will measure the extent to which PEACE Rounds are an effective component on self-help for clinicians and other healthcare workers who care for patients with difficult or controversial treatment plans. Interview questions will include: "What/who do you remember most vividly?" "What was most meaningful to you?" "What would you change about the experience, if you could?" "Would you do it again? Why or why not?" "What, if anything, changed after PEACE rounds?"

CONTACTS AND LOCATIONS:
Overall Officials: Kim S. McManus, Ph.D., Principal Investigator — AdventHealth Center for CREATION Research
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No